CLINICAL TRIAL: NCT04566172
Title: Preoperative Optimization to Improve Functional Status
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to begin the study due to COVID-19 restrictions. Once restrictions were lifted, funding was no longer available.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00227450
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Atelectasis; Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pulmonary Atelectasis; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation program (Experimental): Patient undergoing thoracic or upper abdominal surgery as part of their regular medical care will be approached. Participants will receive a prehabilitation program that includes an inspiratory muscle training that they will do leading up to the day of their surgery.
  Interventions: Behavioral: Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Behavioral: Inspiratory Muscle Training (IMT) — Participants will receive an inspiratory muscle training that they will do leading up to the day of their surgery.
  Other Names: IMT

SUMMARY:
This is a pilot study to obtain preliminary information on the usability and efficacy of a pre-habilitation program. The investigators will recruit up to 100 patients.

The two specific aims of this study are to conduct an initial pilot study with the following goals:

1. To obtain information on feasibility and utilization of the program
2. To determine whether participation in the program improves a patient's Maximal Inspiratory Pressure

DETAILED DESCRIPTION:
Participants will engage in a pre-habilitation program prior to surgery at home, that includes using an inspiratory muscle training (IMT) device that will strengthen the muscles of breathing. Participants will keep a log of training. The Maximum Inspiratory Pressure will be measured at baseline and prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing thoracic or upper abdominal surgery with an estimated date of surgery between 2-10 weeks after enrollment
* Age>65 y/o

Exclusion Criteria:

* Impaired cognition that would limit participation in the program
* History of spontaneous pneumothorax
* Any other physician judgement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Inspiratory muscle training compliance as assessed by daily logs | Up to 10 Weeks
  The primary outcome variable will be compliance with >70% of inspiratory muscle training. Patients will be instructed to follow the prescribed program daily from the day consent is obtained until the day of surgery. Patients will complete a daily log of breathing exercises.

SECONDARY OUTCOMES:
Number of attempted inspiratory muscle training as assessed by percent days the program was attempted | Up to 10 Weeks
  Secondary feasibility outcome variables will be compliance (percent days the program was attempted). Patients will complete a daily log of breathing exercises and document the completion of each breathing exercise. The amount of days to be measured will be the number of days from consent to the day of surgery.
Number of completed inspiratory muscle training as assessed by percent days with full compliance | Up to 10 Weeks
  Secondary feasibility outcome variables will be compliance (percent days with full compliance). Patients will complete a daily log of breathing exercises and document the completion of each breathing exercise. The amount of days to be measured will be the number of days from consent to the day of surgery.
Change in maximum inspiratory pressure | Baseline and on the day of surgery, up to 10 weeks from enrollment
  The change in maximum inspiratory pressure will be determined by comparing the baseline maximum inspiratory pressure to the maximum inspiratory pressure on the day of surgery to assess the efficacy of the inspiratory muscle training.
Interest in Using Program for Future Surgeries as assessed by a likert scale | Day of Surgery, up to 10 weeks from enrollment
  The patient's willingness to use this program for future surgeries will be measured using the Likert scale 1 to 5. Higher scores mean more willingness to use program for future surgeries.
Overall Satisfaction with the Program as assessed by a likert scale | Day of Surgery, up to 10 weeks from enrollment
  The patient's satisfaction with the program will be measure using the Likert scale 1 to 5. Higher scores mean better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brown, MD, Principal Investigator — Johns Hopkins Univesity School of Medicine
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.